CLINICAL TRIAL: NCT02205411
Title: A Prospective, Randomized, Multicenter Clinical Trial to Evaluate the Safety and Efficacy of the HeartAssist 5® VAD System Compared to the Thoratec HeartMate II® VAD and HeartWare® HVAD for Left Ventricular Support in Patients Awaiting Cardiac Transplantation
Brief Title: Clinical Trial to Evaluate the the ReliantHeart HeartAssist 5® VAD System in Patients Awaiting Heart Transplantation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inability to timely enroll.
Sponsor: ReliantHeart Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAP00030
Record Dates: First submitted 2014-07-24; First posted 2014-07-31 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2018-03

CONDITIONS: Heart Failure; Cardiac Failure; Congestive Heart Failure; Heart Failure, Left-sided
Keywords: heart assist device; ventricular assist device
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HeartAssist 5® VAD System (Experimental): Implant of the HeartAssist 5® VAD System
  Interventions: Device: HeartAssist 5® VAD System
- Control VAD (Active Comparator)
  Interventions: Device: Control VAD

INTERVENTIONS:
Device: HeartAssist 5® VAD System — The HeartAssist 5® VAD System is a small, implantable pump that is designed to increase blood flow for patients who have heart failure. The device is intended to support patients in the hospital or at home.
  Arms: HeartAssist 5® VAD System
Device: Control VAD — The HeartMate II® VAD or HVAD®
  Arms: Control VAD

SUMMARY:
The purpose of the study is to evaluate the safety and effectiveness of the ReliantHeart HeartAssist 5® VAD System in patients listed for heart transplantation and at risk of death from refractory end-stage heart failure.

DETAILED DESCRIPTION:
The HeartAssist 5® VAD System is intended for use as a bridge to heart transplantation and will be compared to the HeartMate II and HVAD devices.

Patients that meet the study criteria will be randomized 1:1 to either the HeartAssist 5® VAD System (treatment group) or control group (HeartMate II and HVAD). The physician will have the option to choose which control device to implant.

The primary objective of the study is to show non-inferiority of the HeartAssist 5® (treatment group) to the control group.

ELIGIBILITY:
Inclusion Criteria:

1. Able to sign Informed Consent.
2. Age ≥ 18
3. Body Surface Area (BSA) ≥ 1.2 m2.
4. Cardiac transplant candidate, defined as: Listed for cardiac transplant, and designated by the institution's multidisciplinary transplant committee as appropriate forLVAD Bridge-to-Transplantation therapy, or Designated by the institutions's multidisciplinary transplant committee as: 1) an appropriate candidate for LVAD Bridge-to transplant therapy, and 2) An inappropriate candidate for LVAD destination therapy
5. LVAD implantation has been approved by the institution's multidisciplinary transplant committee.
6. Patient is NYHA Class IV.
7. Able to return to the clinical site for all routine follow up visits.

Exclusion Criteria:

1. Cardiothoracic surgery within 30 days prior to enrollment.
2. Acute Myocardial Infarction within 14 days prior to enrollment.
3. Prior cardiac transplantation, left ventricular reduction surgery, cardiomyoplasty or left ventricular assist device.
4. Mechanical, animal, or human tissue heart valve.
5. History of untreated abdominal or thoracic aortic aneurysm > 5 cm.
6. On ventilator support for > 72 hours within four days immediately prior to enrollment.
7. Ongoing mechanical circulatory support other than an intra-aortic balloon pump (IABP).
8. Proven history of pulmonary embolism within 90 days of enrollment.
9. Moderate to severe aortic insufficiency as determined by echocardiogram without plans for correction during pump implantation surgery.
10. Requires aortic, mitral, tricuspid or pulmonary valve replacements (including Bioprosthetic valves) or left ventricular (LV) aneurysm resection.
11. Uncorrected thrombocytopenia or generalized coagulopathy (e.g., platelets <100,000, INR > 1.6 or PTT > 2.5 times control in the absence of anticoagulation therapy)
12. Severe right ventricular failure as defined by the anticipated need for right ventricular assist device (RVAD) support OR extracorporeal membrane oxygenation (ECMO) at the time of implantation OR right atrial pressure > 20 mmHg while on multiple inotropes.
13. Significant renal dysfunction defined as > 3.5 mg/dl or requires hemo or peritoneal dialysis for renal failure (excluding ultra-filtration for fluid removal).
14. Evidence of intrinsic hepatic disease defined as liver enzyme values (AST, ALT and LDH that are > 3 times the upper limit of normal) OR a total bilirubin > 3 mg/dl OR biopsy proven liver cirrhosis or portal hypertension.
15. Pregnancy
16. Active systemic infection prior to study enrollment not yet resolved by treatment. Active Systemic Infection is defined by any one of the following in spite of antibiotic, antiviral or antifungal treatment: 2 or more consecutive positive cultures; elevated temperature > 37.2 (°C) and white blood cell count > 11.0 (103/ml); hypotension, tachycardia and generalized malaise.
17. Stroke within 90 days prior to enrollment OR patient has a history of cerebral vascular disease with > 80% extra cranial stenosis documented by carotid Doppler study during transplant evaluation
18. Modified Rankin Scale score of ≥ 2 or has any neurologic disability as confirmed by imaging (CT or MRI).
19. Significant lower extremity peripheral vascular disease accompanied by rest pain or leg ulceration.
20. Intolerant to anticoagulant or antiplatelet therapies or any other peri- or postoperative therapy that the investigator may administer based upon the patient's health status.
21. Psychiatric disorder, or other psychosocial behavior that is likely to impair compliance with the study protocol.
22. Receiving therapy with an investigational intervention or participating in any other clinical investigation at the time of enrollment.
23. Condition, other than heart failure, that may limit survival to less than three (3) years and/or would exclude cardiac transplantation.
24. Unwilling or unable to comply with any study requirement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2014-09; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is success at 180 days | 180 days
  Success at 180 days is defined as alive on the original device, transplanted or explanted for heart recovery and alive 60 days after device explant.

SECONDARY OUTCOMES:
Adverse Events | 180 days
  Device safety will be reported as the frequency of each adverse event, (including device failure, device malfunction or unanticipated adverse device effects) and the rate of adverse events per patient year.
Quality of Life | 180 days
  Quality of life data, as measured by the EuroQol (EQ-5D) will be summarized and analyzed, for both groups, comparing data at baseline and study intervals.
Functional Status | 180 days
  NYHA and six-minute walk analysis will be reported by group for data at pre-implant and at study-defined intervals.
Neurologic Status | 180 days
  Evaluation of any change in Modified Rankin Scale from baseline to 180-days post-implant or device explant.

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - University of California San Francisco, San Francisco, California
  - University of Stanford, Stanford, California
  - University of Miami, Coral Gables, Florida
  - University of Chicago Medical Center, Chicago, Illinois
  - Indiana University Health, Inc. d/b/a Methodist Research Institute, Indianapolis, Indiana
  - St. Vincent Hospital & Health Care Center, Indianapolis, Indiana
  - Jewish Hospital, Louisville, Kentucky
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - Mayo Clinic Hospital - Saint Mary's Campus, Rochester, Minnesota
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - CHI St. Luke's Baylor College of Medicine Medical Center, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - University of Texas Health Science Center, Houston, Texas
  - Providence Sacred Heart Hospital, Spokane, Washington